CLINICAL TRIAL: NCT06828016
Title: A Randomized Controlled Study of Foot Reflexology for the Management of Chronic Low Back Pain
Brief Title: Foot Reflexology for Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FJUH112342
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Chronic Low Back Pain; Foot Reflexology
Keywords: chronic low back pain; foot reflexology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-frequency and LBP-focused intervention group (Experimental): foot reflexology, twice weekly, focusing on low back pain, with a total of 12 sessions
  Interventions: Other: foot reflexology
- LBP-focused intervention group (Experimental): foot reflexology, once weekly, focusing on low back pain, with a total of 6 sessions
  Interventions: Other: foot reflexology
- usual care group (Sham Comparator): usual foot care once weekly, primarily for usual foot care, with a total of 6 sessions
  Interventions: Other: usual foot care

INTERVENTIONS:
Other: foot reflexology — foot reflexology, each session lasting 45 minutes to 1 hour
  Arms: High-frequency and LBP-focused intervention group; LBP-focused intervention group
Other: usual foot care — usual foot care, with each session lasting 45 minutes to 1 hour
  Arms: usual care group

SUMMARY:
The aim of this 2-year randomized, double-blinded clinical trial is to investigate the effect of 6 or 12 sessions of weekly 45-minute to 1-hour foot reflexology interventions on physical function and symptoms, pain, health-related quality of life, and ultrasonic shear wave elasticity of plantar fascia among chronic low back pain patients. The results of this study will explore the effect of foot reflexology intervention on physical function and symptoms, pain, health-related quality of life, and ultrasonic shear wave elasticity of plantar fascia among chronic low back pain patients. Our data will also provide relevant scientific evidence and insight into the utility of foot reflexology for the management of chronic low back pain.

DETAILED DESCRIPTION:
Introduction： Foot reflexology is a simple, inexpensive, and non-invasive treatment commonly used to treat various pain problems. The literature review found that Taiwan has not applied clinical trial research methods to evaluate the interventional effectiveness of foot reflexology for chronic low back pain. Therefore, the effect of foot reflexology on chronic low back pain deserves and requires further research.

Objective： The aim of this 2-year randomized, double-blinded clinical trial is to investigate the effect of 6 or 12 sessions of weekly 45-minute to 1-hour foot reflexology interventions on physical function and symptoms, pain, health-related quality of life, and ultrasonic shear wave elasticity of plantar fascia among chronic low back pain patients.

Methods： The patients, 18 years of age or older, with chronic low back pain treated at a regional hospital, will be referred and evaluated for eligibility for the study. The intervention period for foot reflexology is 6-8 weeks, with each session lasting 45 minutes to 1 hour. Participants were divided into three groups using double-blind random assignment based on the level of focus on the low back pain foot reflex zone (LBP-focused) and the frequency of sessions (twice or once per week): the high-frequency and LBP-focused intervention group (twice weekly, focusing on low back pain, with a total of 12 sessions), the LBP-focused intervention group (once weekly, focusing on low back pain, with a total of 6 sessions), and the usual care group (once weekly, primarily for usual foot care, with a total of 6 sessions). The primary outcome was the change in Oswestry Disability Index. The secondary outcome measures include Pain Visual Analogue Scale, Activation Deactivation Adjective Check List, health-related quality of life by Short Form-36, and Shear Wave PLUS Elastography of plantar fascia.

What is New or Innovative in this Study? There is limited evidence regarding efficacy for patients with chronic low back pain undergoing foot reflexology intervention. This prospective randomized, double-blinded, controlled trial will add knowledge regarding foot reflexology for patients with chronic low back pain.

Scientific or Clinical Implication of the Expected Results： The results of this study will explore the effect of foot reflexology intervention on physical function and symptoms, pain, health-related quality of life, and ultrasonic shear wave elasticity of plantar fascia among chronic low back pain patients. Our data will also provide relevant scientific evidence and insight into the utility of foot reflexology for the management of chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain for more than 12 weeks

Exclusion Criteria:

* pregnancy, patients with comorbidities of major injuries or illnesses of National Health Insurance, patients diagnosed with major mental illness according to DSM-V criteria or under the care of mental health services, patients who have had adverse reactions to foot reflexology before, patients with recent surgery or vascular disease of lower extremities, patients who meet contraindications to foot reflexology.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | From enrollment to the end of treatment at 12 week
  The change of Oswestry Disability Index

SECONDARY OUTCOMES:
Pain Visual Analogue Scale | From enrollment to the end of treatment at 12 week
  The change of Pain Visual Analogue Scale
Activation Deactivation Adjective Check List | From enrollment to the end of treatment at 12 week
  The change of Activation Deactivation Adjective Check List
Health-related quality of life by Short Form-36 | From enrollment to the end of treatment at 12 week
  The change of health-related quality of life by Short Form-36
Shear wave elastography of plantar fascia | From enrollment to the end of treatment at 12 week
  The change of shear wave elastography of plantar fascia

CONTACTS AND LOCATIONS:
Overall Officials: Ssu-Yuan Chen, MD, PhD,, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No